CLINICAL TRIAL: NCT02550769
Title: Multicenter Prospective Randomized Controlled Study of the Transanal Total Mesorectal Excision Versus Laparoscopic Low Anterior Resection in Rectal Cancer
Brief Title: Study of NOTES-TME Versus L-LAR in Rectal Cancer
Acronym: NOTESvsL-LAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Xavier Serra-Aracil, Medical Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOTES-LRAB_TAU-2015
Record Dates: First submitted 2015-08-31; First posted 2015-09-16 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2020-07

CONDITIONS: Rectal Cancer
Keywords: Transanal NOTES; Transanal TME; Laparoscopic Low Anterior Resection; Surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRANSANAL TOTAL MESORECTAL EXCISION (Experimental): Transanal approach of total mesorectal excision.
  Interventions: Procedure: TRANSANAL TOTAL MESORECTAL EXCISION
- Laparoscopic-LAR (Active Comparator): Type of surgical intervention as control group: Laparoscopic low anterior resection with total mesorectal excision for rectal cancer
  Interventions: Procedure: Laparoscopic-LAR

INTERVENTIONS:
Procedure: TRANSANAL TOTAL MESORECTAL EXCISION — The technique begins with the TEO equipment and a purse string 1 cm distal to the tumor. The dissection progresses in the posterior part until the laparoscopic TME field is reached. After the section of the rectum and TME transanal dissection, the anvil of the circular mechanical stapler is introduced through the TEO rectoscope. In the laparoscopic field, the mesosigma is sectioned at the point where the colon section is to be performed. The TEO rectoscope is withdrawn, and the bag containing the specimen is removed through the anus. The stapler is inserted. From the laparoscopic field, the strings of the purse are tightened and the purse is closed around the rectal stump with a clip. Then the stapler are joined to perform the anastomosis and a loop ileostomy is placed in the right flank.
  Arms: TRANSANAL TOTAL MESORECTAL EXCISION
Procedure: Laparoscopic-LAR — Standard laparoscopic low anterior resection of the rectum with total mesorectal excision and colorectal anastomosis
  Other Names: Laparoscopic Low Anterior Resecion of the rectum
  Arms: Laparoscopic-LAR

SUMMARY:
INTRODUCTION: Transanal TME (T-TME) combined with laparoscopy, called hybrid-NOTES, is a less invasive procedure that responds to some of the limitations of the rectal laparoscopic approach.

MAIN OBJECTIVE: To analyze that the T-TME gets a faster recovery due to a lower conversion rate to open surgery than laparoscopic low anterior resection (L-LAR) in rectal cancer with the same pathological, functional and oncologic results.

METHODOLOGY: A prospective multicenter randomized controlled study of patients with rectal cancer that, were randomized in the T-TME- and L-LAR group. The main variables are: general morbidity, anastomotic dehiscence, conversion rate to open surgery and hospital stay. The sample calculation is 58 patients per group.

DETAILED DESCRIPTION:
INTRODUCTION: The laparoscopic total mesorectal excision (TME) has provided better patient recovery with less morbidity and shorter hospital stay compared with open surgery. However in laparoscopic low rectal surgery, overall conversion to open surgery is around 20%. Transanal TME (T-TME) combined with laparoscopy, called hybrid-NOTES, is a less invasive procedure that responds to some of the limitations of the rectal laparoscopic approach.

MAIN OBJECTIVE: To analyze that the T-TME gets a faster recovery due to a lower conversion rate to open surgery than laparoscopic low anterior resection (L-LAR) in rectal cancer with the same pathological, functional and oncologic results.

METHODOLOGY: A prospective multicenter randomized controlled study of patients diagnosed with adenocarcinoma of the rectum that after inclusion and exclusion criteria, were randomized in the T-TME- and L-LAR group. The main variables are: general morbidity, anastomotic dehiscence, conversion rate to open surgery and hospital stay. The other variables studied were: demographic, surgical, pathological, 30-day morbidity and mortality, quality of life and oncologic results. The sample calculation is 53 patients per group. With an estimated loss of 10%, the final number will be 116 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients with rectal cancer stage: cT1-2-3, cN0-1, cM0.
* Tumor equal or below 10 cm from the anal verge, candidates to (ETM) low anterior resection and anastomosis, with or without preoperative chemo-radiotherapy.
* Adenocarcinoma of low or moderate differentiation
* ASA I, II, III.

Exclusion Criteria:

* Do not sign informed consent
* Pregnant patients
* Liver cirrhosis
* Undifferentiated adenocarcinoma.
* cT4
* Metastatic disease (M1)
* chronic renal failure on dialysis
* ASA IV
* BMI <18 and> 35 kg / m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the T-TME versus L-LAR with the Dindo-Claviens classification in patients with rectal cancer. | 30 days
  Evaluate surgical complications 30 days after surgery.
Evaluate the effectiveness of the T-TME versus L-LAR with the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) CR-30 score in patients with rectal cancer. | 6 months
  Evaluate functional results 6 months after ileostomy closure.
Evaluate the effectiveness of the T-TME versus L-LAR with the EORTC QLQ-CR29 score in patients with rectal cancer. | 6 months
  Evaluate functional results 6 months after ileostomy closure.
Evaluate the effectiveness of the T-TME versus L-LAR with the LARS score in patients with rectal cancer. | 6 months
  Evaluate functional results 6 months after ileostomy closure.

CONTACTS AND LOCATIONS:
Overall Officials: Serra-Aracil Xavier, MD, PhD, Principal Investigator — Corporacio Parc Tauli. Parc Tauli University Hospital
Locations (1):
- Parc Tauli University Hospital, Sabadell, Barcelona, Spain

REFERENCES:
- [Background] Serra-Aracil X, Mora-Lopez L, Casalots A, Pericay C, Guerrero R, Navarro-Soto S. Hybrid NOTES: TEO for transanal total mesorectal excision: intracorporeal resection and anastomosis. Surg Endosc. 2016 Jan;30(1):346-54. doi: 10.1007/s00464-015-4170-5. Epub 2015 Mar 27. PMID 25814073
- [Background] Serra-Aracil X. [Transanal total mesorectal excision]. Cir Esp. 2014 Apr;92(4):221-2. doi: 10.1016/j.ciresp.2014.01.002. Epub 2014 Feb 24. No abstract available. Spanish. PMID 24576748
- [Derived] Serra-Aracil X, Zarate A, Bargallo J, Gonzalez A, Serracant A, Roura J, Delgado S, Mora-Lopez L; Ta-LaTME study Group. Transanal versus laparoscopic total mesorectal excision for mid and low rectal cancer (Ta-LaTME study): multicentre, randomized, open-label trial. Br J Surg. 2023 Jan 10;110(2):150-158. doi: 10.1093/bjs/znac324. PMID 36224406
- [Derived] Serra-Aracil X, Zarate A, Mora L, Serra-Pla S, Pallisera A, Bonfill J, Bargallo J, Pando A, Delgado S, Balleteros E, Pericay C. Study protocol for a multicenter prospective controlled and randomized trial of transanal total mesorectal excision versus laparoscopic low anterior resection in rectal cancer. Int J Colorectal Dis. 2018 May;33(5):649-655. doi: 10.1007/s00384-018-2996-8. Epub 2018 Mar 16. PMID 29546560